CLINICAL TRIAL: NCT07258823
Title: Study on the Effectiveness of Continuous Compression-synchronous Ventilation (Bio-CPR) in the ACLS Stage of Cardiopulmonary Resuscitation (ACLS) Based on the Bionic Concept to Explore the Best Mechanical Ventilation Strategy
Brief Title: the Effectiveness of Continuous Compression-synchronous Ventilation (Bio-CPR)
Acronym: Bio-CPR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, lixin, Vice President, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ChiCTR2400094466
Record Dates: First submitted 2025-11-21; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Out-of-hospital Cardiac Arrest (OHCA); Cardiac Arrest (CA); CPR; ACLS
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest | interventions — Cardiopulmonary Resuscitation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bio-CPR experimental group (Experimental): Bio-CPR ventilation mode
  Interventions: Procedure: CPR
- Traditional compression/ventilation mode group (Active Comparator): Traditional compression/ventilation mode
  Interventions: Procedure: CPR

INTERVENTIONS:
Procedure: CPR — ACLS/CPR (Bio-CPR Group vs. Traditional Resuscitation Group)
  This intervention targets adult patients with in-hospital or out-of-hospital cardiac arrest (CA) who require advanced resuscitation. All patients receive immediate basic life support (BLS) upon medical contact, followed by standardized advanced cardiac life support (ACLS) with uniform use of the integrated "CPR Machine E8 - Ventilator T7" system (distinguishing it from manual CPR or other device-based protocols). Randomization determines two subgroups with distinct ventilation and compression-coordination settings, as detailed below:
  1. Core Uniform Foundation (Applicable to Both Groups) Chest Compression Mode: Continuous compression mode is activated on the CPR Machine E8, eliminating variability from manual compression rate/depth and ensuring consistent compression quality.
  Airway & Vascular Access: Advanced airway (e.g., endotracheal intubation) is established as soon as possible post-BLS initiation; peripheral or central

SUMMARY:
Bio-CPR is an innovative new mechanical resuscitation model proposed by our research group. A multi-center RCT study was established to comprehensively evaluate the efficacy of this model and the current standard CPR protocol, verify its safety and efficacy, and provide high-quality clinical evidence support.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years old; 2. Cardiac arrest with witnesses; 3. Onset - compression start time<5 minutes; 4. Initial ventricular fibrillation rhythm; 5. Endotracheal intubation and use of a mechanical chest CPR device; Patients with OHCA who meet the above conditions

Exclusion Criteria:

* 1. OHCA patients who are not suitable for mechanical compression ventilation; 2. The participant or his/her legally authorized representative (LAR) is unable or unwilling to provide written informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Mean tidal volume | 15 minutes
  Mean tidal volume

SECONDARY OUTCOMES:
Mean minute ventilation and end-tidal carbon dioxide | 15 minutes
  Ventilation monitoring: EtCO2, dynamic monitoring of ventilator mechanical parameters, PEEPi+P0.1, tidal volume and minute ventilation volume were selected as the quality index of ventilation, and end-expiratory carbon dioxide was selected as the quality index of gas exchange. These values are collected by the ventilator software.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kamler M, Lehr HA, Barker JH, Saetzler RK, Galla TJ, Messmer K. Impact of ischemia on tissue oxygenation and wound healing: intravital microscopic studies on the hairless mouse ear model. Eur Surg Res. 1993 Jan-Feb;25(1):30-7. doi: 10.1159/000129254. PMID 8482303
- [Result] Greif R, Bray JE, Djarv T, Drennan IR, Liley HG, Ng KC, Cheng A, Douma MJ, Scholefield BR, Smyth M, Weiner G, Abelairas-Gomez C, Acworth J, Anderson N, Atkins DL, Berry DC, Bhanji F, Bottiger BW, Bradley RN, Breckwoldt J, Carlson JN, Cassan P, Chang WT, Charlton NP, Phil Chung S, Considine J, Cortegiani A, Costa-Nobre DT, Couper K, Couto TB, Dainty KN, Dassanayake V, Davis PG, Dawson JA, de Caen AR, Deakin CD, Debaty G, Del Castillo J, Dewan M, Dicker B, Djakow J, Donoghue AJ, Eastwood K, El-Naggar W, Escalante-Kanashiro R, Fabres J, Farquharson B, Fawke J, de Almeida MF, Fernando SM, Finan E, Finn J, Flores GE, Foglia EE, Folke F, Goolsby CA, Granfeldt A, Guerguerian AM, Guinsburg R, Hansen CM, Hatanaka T, Hirsch KG, Holmberg MJ, Hooper S, Hoover AV, Hsieh MJ, Ikeyama T, Isayama T, Johnson NJ, Josephsen J, Katheria A, Kawakami MD, Kleinman M, Kloeck D, Ko YC, Kudenchuk P, Kule A, Kurosawa H, Laermans J, Lagina A, Lauridsen KG, Lavonas EJ, Lee HC, Han Lim S, Lin Y, Lockey AS, Lopez-Herce J, Lukas G, Macneil F, Maconochie IK, Madar J, Martinez-Mejas A, Masterson S, Matsuyama T, Mausling R, McKinlay CJD, Meyran D, Montgomery W, Morley PT, Morrison LJ, Moskowitz AL, Myburgh M, Nabecker S, Nadkarni V, Nakwa F, Nation KJ, Nehme Z, Nicholson T, Nikolaou N, Nishiyama C, Norii T, Nuthall G, Ohshimo S, Olasveengen T, Olaussen A, Ong G, Orkin A, Parr MJ, Perkins GD, Pocock H, Rabi Y, Raffay V, Raitt J, Raymond T, Ristagno G, Rodriguez-Nunez A, Rossano J, Rudiger M, Sandroni C, Sawyer TL, Schexnayder SM, Schmolzer G, Schnaubelt S, Seidler AL, Semeraro F, Singletary EM, Skrifvars MB, Smith CM, Soar J, Solevag AL, Soll R, Stassen W, Sugiura T, Thilakasiri K, Tijssen J, Tiwari LK, Topjian A, Trevisanuto D, Vaillancourt C, Welsford M, Wyckoff MH, Yang CW, Yeung J, Zelop CM, Zideman DA, Nolan JP, Berg KM. 2024 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations: Summary From the Basic Life Support; Advanced Life Support; Pediatric Life Support; Neonatal Life Support; Education, Implementation, and Teams; and First Aid Task Forces. Circulation. 2024 Dec 10;150(24):e580-e687. doi: 10.1161/CIR.0000000000001288. Epub 2024 Nov 14. PMID 39540293
- [Result] Berg KM, Soar J, Andersen LW, Bottiger BW, Cacciola S, Callaway CW, Couper K, Cronberg T, D'Arrigo S, Deakin CD, Donnino MW, Drennan IR, Granfeldt A, Hoedemaekers CWE, Holmberg MJ, Hsu CH, Kamps M, Musiol S, Nation KJ, Neumar RW, Nicholson T, O'Neil BJ, Otto Q, de Paiva EF, Parr MJA, Reynolds JC, Sandroni C, Scholefield BR, Skrifvars MB, Wang TL, Wetsch WA, Yeung J, Morley PT, Morrison LJ, Welsford M, Hazinski MF, Nolan JP; Adult Advanced Life Support Collaborators. Adult Advanced Life Support: 2020 International Consensus on Cardiopulmonary Resuscitation and Emergency Cardiovascular Care Science With Treatment Recommendations. Circulation. 2020 Oct 20;142(16_suppl_1):S92-S139. doi: 10.1161/CIR.0000000000000893. Epub 2020 Oct 21. PMID 33084390
- [Result] Nichol G, Leroux B, Wang H, Callaway CW, Sopko G, Weisfeldt M, Stiell I, Morrison LJ, Aufderheide TP, Cheskes S, Christenson J, Kudenchuk P, Vaillancourt C, Rea TD, Idris AH, Colella R, Isaacs M, Straight R, Stephens S, Richardson J, Condle J, Schmicker RH, Egan D, May S, Ornato JP; ROC Investigators. Trial of Continuous or Interrupted Chest Compressions during CPR. N Engl J Med. 2015 Dec 3;373(23):2203-14. doi: 10.1056/NEJMoa1509139. Epub 2015 Nov 9. PMID 26550795
- [Result] Zheng J, Lv C, Zheng W, Zhang G, Tan H, Ma Y, Zhu Y, Li C, Han X, Yan S, Pan C, Zhang J, Hou Y, Wang C, Bian Y, Liu R, Cheng K, Ma J, Zheng Z, Song R, Wang M, Gu J, McNally B, Ong MEH, Chen Y, Xu F; BASIC-OHCA Coordinators and Investigators. Incidence, process of care, and outcomes of out-of-hospital cardiac arrest in China: a prospective study of the BASIC-OHCA registry. Lancet Public Health. 2023 Dec;8(12):e923-e932. doi: 10.1016/S2468-2667(23)00173-1. Epub 2023 Sep 16. PMID 37722403
- [Result] Nichols JH, Howard C, Loman K, Miller C, Nyberg D, Chan DW. Laboratory and bedside evaluation of portable glucose meters. Am J Clin Pathol. 1995 Feb;103(2):244-51. doi: 10.1093/ajcp/103.2.244. PMID 7856571
- [Result] Panchal AR, Bartos JA, Cabanas JG, Donnino MW, Drennan IR, Hirsch KG, Kudenchuk PJ, Kurz MC, Lavonas EJ, Morley PT, O'Neil BJ, Peberdy MA, Rittenberger JC, Rodriguez AJ, Sawyer KN, Berg KM; Adult Basic and Advanced Life Support Writing Group. Part 3: Adult Basic and Advanced Life Support: 2020 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2020 Oct 20;142(16_suppl_2):S366-S468. doi: 10.1161/CIR.0000000000000916. Epub 2020 Oct 21. No abstract available. PMID 33081529
- [Result] Schmidt H, Kjaergaard J, Hassager C, Molstrom S, Grand J, Borregaard B, Roelsgaard Obling LE, Veno S, Sarkisian L, Mamaev D, Jensen LO, Nyholm B, Hofsten DE, Josiassen J, Thomsen JH, Thune JJ, Lindholm MG, Stengaard Meyer MA, Winther-Jensen M, Sorensen M, Frydland M, Beske RP, Frikke-Schmidt R, Wiberg S, Boesgaard S, Lind Jorgensen V, Moller JE. Oxygen Targets in Comatose Survivors of Cardiac Arrest. N Engl J Med. 2022 Oct 20;387(16):1467-1476. doi: 10.1056/NEJMoa2208686. Epub 2022 Aug 27. PMID 36027567
- [Result] Fuest K, Dorfhuber F, Lorenz M, von Dincklage F, Morgeli R, Kuhn KF, Jungwirth B, Kanz KG, Blobner M, Schaller SJ. Comparison of volume-controlled, pressure-controlled, and chest compression-induced ventilation during cardiopulmonary resuscitation with an automated mechanical chest compression device: A randomized clinical pilot study. Resuscitation. 2021 Sep;166:85-92. doi: 10.1016/j.resuscitation.2021.07.010. Epub 2021 Jul 22. PMID 34302927
- [Result] van Eijk JA, Doeleman LC, Loer SA, Koster RW, van Schuppen H, Schober P. Ventilation during cardiopulmonary resuscitation: A narrative review. Resuscitation. 2024 Oct;203:110366. doi: 10.1016/j.resuscitation.2024.110366. Epub 2024 Aug 23. PMID 39181499
- [Result] Tang Y, Sun M, Zhu A. Outcome of cardiopulmonary resuscitation with different ventilation modes in adults: A meta-analysis. Am J Emerg Med. 2022 Jul;57:60-69. doi: 10.1016/j.ajem.2022.04.027. Epub 2022 Apr 27. PMID 35525159
- [Result] Richman CM, Makii MM, Weiser PA, Herbst AL. The effect of lithium carbonate on chemotherapy-induced neutropenia and thrombocytopenia. Am J Hematol. 1984 May;16(4):313-23. doi: 10.1002/ajh.2830160402. PMID 6426295
- [Result] Zussman L, Zussman S, Sunley R, Bjornson E. Sexual response after hysterectomy-oophorectomy: recent studies and reconsideration of psychogenesis. Am J Obstet Gynecol. 1981 Aug 1;140(7):725-9. doi: 10.1016/0002-9378(81)90730-4. PMID 7196155
- [Result] Suverein MM, Delnoij TSR, Lorusso R, Brandon Bravo Bruinsma GJ, Otterspoor L, Elzo Kraemer CV, Vlaar APJ, van der Heijden JJ, Scholten E, den Uil C, Jansen T, van den Bogaard B, Kuijpers M, Lam KY, Montero Cabezas JM, Driessen AHG, Rittersma SZH, Heijnen BG, Dos Reis Miranda D, Bleeker G, de Metz J, Hermanides RS, Lopez Matta J, Eberl S, Donker DW, van Thiel RJ, Akin S, van Meer O, Henriques J, Bokhoven KC, Mandigers L, Bunge JJH, Bol ME, Winkens B, Essers B, Weerwind PW, Maessen JG, van de Poll MCG. Early Extracorporeal CPR for Refractory Out-of-Hospital Cardiac Arrest. N Engl J Med. 2023 Jan 26;388(4):299-309. doi: 10.1056/NEJMoa2204511. PMID 36720132
- [Result] Robinson H. Make phosphorus education hit home! J Ren Nutr. 1998 Jan;8(1):46-7. doi: 10.1016/s1051-2276(98)90038-3. No abstract available. PMID 9724830